CLINICAL TRIAL: NCT02044484
Title: HIV Clinic-Based Intervention to Improve ART Adherence and Prevent HIV Transmission
Acronym: APTcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-2468; CDC (Other: CDC)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: HIV; AIDS; Viral load; Primary care
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-component intervention (Experimental): Computer-based intervention (CBI) completed twice (separated by 2-4 months) among patients whose viral load exceeds 1000 copies/mL at time of enrollment.
  One-on-one counseling from a project Health Coach (three 1-hour sessions at the clinic and two follow-up phone calls at 1 and 3 months after last session). The counseling is offered to patients who do not show a 1-log reduction in their viral load after the first CBI or whose viral load remains above 200 copies/mL after two administrations of the CBI.
  Behavioral screening of patients at HIV primary care visits.
  Dissemination of palm cards with empowering messages at HIV primary care visits.
  Interventions: Behavioral: Multi-component intervention
- Standard of care control (No Intervention): HIV patients will continue to receive existing standard of care practices at the clinic without receiving the multi-component intervention.

INTERVENTIONS:
Behavioral: Multi-component intervention — The computer-based intervention (CBI) is offered to patients whose viral load exceeds 1000 copies/mL at enrollment.
  Counseling is offered to patients whose viral load does not drop 1-log after the first CBI or remains above 200 copies/mL after completing two CBIs.
  The behavioral screener will be conducted of all patients at primary care visits. The patient completes the screener before seeing the provider. Responses are given to their provider who can use it in clinical care of the patient.
  At primary care visits, all patients are given a palm card containing 1 of 15 empowering messages before they leave the clinic. Messages cover three domains: adhering to antiretroviral therapy, regular care, and safer sex.
  Arms: Multi-component intervention

SUMMARY:
This research, co-sponsored by the Centers for Disease Control and Prevention and the National Institute of Mental health, is conducted at six HIV clinics in the U.S. The research examines the effect of a clinic-based multi-component intervention delivered to HIV patients when they attend clinic for primary care. The study tests the hypothesis that the intervention will improve the viral load status of patients and improve attendance for HIV primary care.

DETAILED DESCRIPTION:
This study examines the effect of an HIV clinic-based multi-component intervention on HIV patients' subsequent viral load status and attendance for HIV primary care. The intervention has clinic-wide and targeted components. The clinic-wide components are given to all HIV patients when they attend clinic for primary care and include: (1) patient behavioral screening used by providers in the clinical care of patients and (2) dissemination of palm cards which contain messages about the importance of adhering to antiretroviral therapy (ART), coming to clinic regularly, and safer sex. The targeted components focus on patients whose viral loads exceed 1000 copies/mL. Targeted components include: (1) an interactive computer-based intervention (CBI) completed twice (separated by 2-4 months) by patients at the clinic and (2) referral for one-on-one counseling from trained project Health Coaches if the patient's viral load does not show a 1-log reduction after the first CBI or remains above 200 copies/mL after two administrations of the CBI.

Patients are not individually randomly assigned to arms. The multi-component intervention is evaluated using a group-randomized design. Clinics were randomized to either Panel A or Panel B with the intent of equating the two panels on the percentage of patients with suppressed viral load prior to implementing the intervention. Three clinics (Panel A) begin intervention activities, and the other three clinics (Panel B) delay onset of all intervention activities for 16 months and thus serve as a concurrent control group during that 16-month period. This enables between-panel comparisons of the outcomes during this time interval.

The primary analytic cohort for the group-randomized analysis will be all patients in Panel A and Panel B whose viral load exceeds 1000 copies/mL who have a scheduled primary care appointment during a 7-month enrollment period. Viral load eligible patients in Panel A will be part of the analytic cohort regardless of whether they enroll in the CBI or not. These viral load eligible patients represent the group of patients who are targeted for the main intervention components (CBI and counseling) and, accordingly, will comprise the denominator (estimated to be 2,794) for the primary analysis of the viral load and clinic attendance outcomes. Each cohort member in Panel A is followed for 9 months for purpose of delivering the intervention and assessing the outcomes. Each cohort member in Panel B is followed for 9 months for purpose of assessing the outcomes.

Two secondary levels of analysis will also be performed. First, analysis will be performed focusing on all patients in Panel A clinics who have a viral load over 1000 copies/mL and received at least one administration of the CBI ("as-treated" approach). Outcomes of these patients will be compared to patients in Panel B whose viral load exceeds 1000 copies/mL during the recruitment period. Second, an analysis will be performed at the clinic-wide level including all patients in Panel A clinics regardless of viral load level who are scheduled for primary care during the recruitment period. Outcomes of these patients will be compared to all patients in Panel B scheduled for primary care visits during the recruitment period.

ELIGIBILITY:
Inclusion Criteria:

* All patients are eligible to receive behavioral screening and palm cards
* Patients with viral load exceeding 1000 copies/mL are eligible for the computer-based intervention and referral to counseling

Exclusion Criteria:

* Patients under the age of 18 (under 19 in Alabama) are not eligible for the computer-based intervention or referral to counseling because they cannot provide legal informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2794 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with suppressed HIV (≤ 200 copies/mL) | At 9-month time point
Percentage of patients without a gap in HIV primary care (without a gap > 6 months) | From baseline to 9-month time point

SECONDARY OUTCOMES:
Change across time in log10 viral load values | From baseline to 9-month time point
HIV primary care appointment adherence | From baseline to 9-month time point
  Proportion of scheduled HIV primary care appointments kept (omitting prior cancellations) per patient

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Giordano, MD, Principal Investigator — Baylor College of Medicine; Margaret Sullivan, MD, Principal Investigator — Boston University; Matthew Golden, MD, Principal Investigator — University of Washington; Edward Cachay, MD, Principal Investigator — University of California, San Diego; Michael J Mugavero, MD, Principal Investigator — University of Alabama at Birmingham; Allan E Rodriguez, MD, Principal Investigator — University of Miami
Locations (6):
- United States (6):
  - 1917 Clinic, Birmingham, Alabama
  - Owen Clinic, San Diego, California
  - Jackson Memorial Hospital, Miami, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Thomas Street Health Center, Houston, Texas
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Stirratt MJ, Marks G, O'Daniels C, Cachay ER, Sullivan M, Mugavero MJ, Dhanireddy S, Rodriguez AE, Giordano TP. Characterising HIV transmission risk among US patients with HIV in care: a cross-sectional study of sexual risk behaviour among individuals with viral load above 1500 copies/mL. Sex Transm Infect. 2018 May;94(3):206-211. doi: 10.1136/sextrans-2017-053178. Epub 2017 Nov 2. PMID 29097417